CLINICAL TRIAL: NCT01541176
Title: Impact of the Absence of Steroids on the Evolution of Renal Function and on the Progression of Graft Fibrosis, Quantified by Numerical Method, in Patients With Renal Transplant
Brief Title: Absence of Steroid in Renal Transplantation and Digital Fibrosis Observation
Acronym: Astronef
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC11_0013
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Renal Transplant
Keywords: Corticotherapy; Fibrosis; Numerical reading; 18-70 years; first renal transplant was lost due to rejection; first or second renal transplant
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absence of corticotherapy post-transplantation (Experimental): All patients included in this arm will receive the usual treatment strategy (including Advagraf, Cellcept ou Myfortic and Simulect) without corticotherapy post-transplantation.
  Interventions: Other: Absence of corticotherapy post-transplantation
- Corticotherapy post-transplantation (Active Comparator): All patients included in this arm will receive the usual treatment strategy (including Advagraf, Cellcept ou Myfortic and Simulect) with corticotherapy post-transplantation : prednisone or prednisolone orally for at least one year post-transplantation.
  Interventions: Drug: Corticotherapy post-transplantation

INTERVENTIONS:
Other: Absence of corticotherapy post-transplantation — No study treatment
  Arms: Absence of corticotherapy post-transplantation
Drug: Corticotherapy post-transplantation — Prednisone or prednisolone orally for at least one year post-transplantation with the following minimal doses :
  * D1 to D14 : 20 mg/day,
  * D15 to M1 : 15 mg/day,
  * M1 to M3 : 10 mg/day,
  * M3 to M12 : 5 mg/day.
  Arms: Corticotherapy post-transplantation

SUMMARY:
The main objective of this study is to demonstrate that the absence of post-transplantation corticosteroids does not induce a larger increase of renal graft fibrosis (by numerical reading) on biopsy at one year post-transplantation than immunosuppressive treatment strategy that includes standard oral corticosteroids.The secondary objectives of the study consist to compare on various parameters (fibrosis progression, renal function, dialysis, ratio of proteinuria/creatinuria, acute rejection, donor-specific antibody, graft survival, clinical and biological tolerance) therapy with no corticosteroids post-transplantation in comparison to standard immunosuppressive treatment strategies including oral corticosteroids. Secondary objectives of the study consist also to compare the two techniques for assessing fibrosis by numerical reading and by centralized blinded reading of the treatment group (by 2 anatomical pathologists).

ELIGIBILITY:
Pre-Inclusion Criteria:

* Adults aged 18 to70 years,
* Accepting to give, after information, their signed informed consent form,
* Not having difficulties to understand and communicate with the investigator and his representatives,
* Requiring a renal transplant [first or second transplant (except if the first renal transplant was lost due to rejection)],
* Patient insured.

Inclusion criteria :

* Transplant of a kidney from a deceased or living donor (non HLA-identical) with ABO compatibility,
* Existence of a renal graft biopsy (or of one of the grafts, if bi-renal transplant) before transplantation,
* Percentage of positive responses to PRA (panel reactive antibodies), measured by the Luminex® less than 20% of IgG anti-T or absence of positive DSA by Luminex regardless of the mean fluorescence (MFI) within the last 6 months,
* Negative cross match T in cytotoxicity and / or flow cytometry,
* Negative pregnancy test for patients of childbearing age, and consent to use an effective contraception throughout the study and 6 weeks after the end of the study.

Exclusion Criteria:

* First renal transplant lost due to rejection,
* Combined transplantation,
* Previous history of transplantation other than kidney,
* Non beating donor heart,
* Presence of positive DSA by Luminex® regardless of the average of fluorescence (MFI),
* Patients receiving corticosteroids at the time of transplantation,
* Necessity to continue administration of systemic immunosuppressive treatment before transplantation,
* Infections or severe diarrhea, vomiting, upper gastrointestinal tract malabsorption or active peptic ulcers, concomitant, significant and uncontrolled,
* Subject or HIV positive donor,
* Replicating viral hepatitis at the time of randomization,
* Known allergy or intolerance to tacrolimus, macrolide, corticosteroids, mycophenolate mofetil or to any of the excipients,
* Diagnosis of de novo malignancy prior to transplantation, with the exception of treated effectively basal cell or squamous cell carcinomas of the skin,- Current participation at another clinical study,
* All clinical condition that the investigator considers incompatible with the conduct of the study in acceptable security conditions,
* Inability of patient to comply with study procedures,
* Pregnant or breast-feeding women,
* Person placed under guardianship, under protection of law.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Percentage of fibrosis of the graft | One year post-transplantation
  Evolution of the percentage of fibrosis of the graft during the first year after transplantation (pre-transplant biopsy versus biopsy at one year), by numerical reading of fibrosis by image analysis.

SECONDARY OUTCOMES:
Percentage of fibrosis of the graft | One year post-transplantation
  Evolution of the percentage of fibrosis of the graft during the first year after transplantation (pre-transplant biopsy versus biopsy at one year of which the blinded readings to treatment group are made by two independent anatomical pathologists, the Banff criteria 2009).
Percentage of fibrosis of the graft. | One year post-transplantation
  The percentage of fibrosis of the graft at one year post-transplantation (biopsy at one year with numerical reading of fibrosis by image analysis and blinded reading to treatment group by two independent anatomical pathologists, the Banff criteria 2009).
Average glomerular filtration rate | One year post-transplantation
  The average glomerular filtration rate, calculated by the MDRD formula (four variables, Modification Diet in Renal Disease).
Dialysis session | One year post-transplantation
  The percentage of patients with at least one dialysis session realised during the first year of transplant.
Ratio of proteinuria/creatinuria | One year post-transplantation
  Average of ratio of proteinuria/creatininuria (mg / mmol).
Episode of acute rejection | One year post-transplantation
  The percentage of patients with at least one episode of acute rejection during the first year after transplantation. We will distinguish biopsy-proven acute rejection (RABP), the corticosteroids resistant RABP and severe RABP (Banff 2009).
Diagnosis of DSA | One year post-transplantation
  The percentage of patients with a diagnosis of DSA (Luminex® method) at 3 months and 1 year post-transplantation.
Percentage of graft failure | One year post-transplantation
  The percentage of graft failure (death or return to dialysis) during the first year of transplantation (the short duration of the study avoids the management of right censoring).
Difference between numerical reading of fibrosis and evaluation by anatomical pathologists | One year post-transplantation
  The difference between the percentage of graft fibrosis evaluated by numerical reading of fibrosis and that assessed by two independent anatomical pathologists (Banff 2009 criteria) at baseline, 3 months and 1 year post-transplantation.
Number of adverse events | One year post-transplantation
  Adverse events (AE) at 12 months post-transplantation, of which AEs of special interest (NODAT, dyslipidemia, hypertension, CMV viral infections, BKV) with an assessment of vital signs, physical examinations and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Diego CANTAROVICH, MD, PhD, Principal Investigator — Nantes University Hospital; Lionel ROSTAING, Profesor, Study Chair — University Hospital, Toulouse; Christophe LEGENDRE, Profesor, Study Chair — Hôpital Necker (AP-HP); Emmanuel MORELON, Profesor, Study Chair — Hospices Civils de Lyon; Elisabeth CASSUTO-VIGUIER, Doctor, Study Chair — Centre Hospitalier Universitaire de Nice; Christophe MARIAT, Profesor, Study Chair — CHU de Saint-Etienne; Matthias BÜCHLER, Profesor, Study Chair — CHRU de Tours; Antoine DURRBACH, Profesor, Study Chair — Hôpital Bicêtre (AP-HP)
Locations (8):
- France (8):
  - CHU de Lyon, Lyon
  - Nantes University Hospital, Nantes
  - CHU de Nice, Nice
  - AP-HP - Hôpital Necker, Paris
  - AP-HP - Hôpital Bicêtre, Paris
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours